CLINICAL TRIAL: NCT04277026
Title: Mindfulness Training for Adults With Physical Inactivity
Brief Title: Mindful Walking Intervention for Physical Inactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: YMCA (Other); Prisma Health-Upstate (Other)
Responsible Party: Principal Investigator, Heidi Zinzow, Associate Professor, Clemson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00092710
Record Dates: First submitted 2020-02-14; First posted 2020-02-20 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with a waitlist control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Walking (Experimental): Eight weekly 60 minute mindful walking sessions involving observations of bodily sensations, experiences, and breath. Discussion of mindful walking experiences and encouragement to meet physical activity goals. The intervention will take place two times per week for four weeks (Weeks 1-4). During weeks 5-8 the experimental group will continue treatment as usual and will not be receiving the mindful walking intervention.
  Interventions: Behavioral: Mindful Walking
- Control (No Intervention): Participants will engage in treatment as usual during the first four weeks and will not be receiving the experimental intervention (mindful walking) during weeks 1-4. After the experimental group completes the mindful walking intervention, the control group will complete the mindful walking intervention (weeks 5-8).

INTERVENTIONS:
Behavioral: Mindful Walking — Eight weekly 60 minute mindful walking sessions involving observations of bodily sensations, experiences, and breath. Discussion of mindful walking experiences and encouragement to meet physical activity goals.
  Arms: Mindful Walking

SUMMARY:
Mindful walking is a meditation practice that combines physical activity and mindfulness practice. The purpose of this study is to examine the effectiveness of mindfulness-based interventions provided for increasing physical activity among adults with low physical activity levels. A randomized controlled trial design will be utilized, with an intervention and waitlist control group (N = 160). Outcomes measured include physical activity, sleep quality, and functional fitness. Participants will receive a total of eight sessions of 60-minute mindful walking training within four weeks. The intervention group will receive the training in Weeks 1-4 and the control group will receive the training during Weeks 5-8. Each training group will consist of up to 20 individuals. Data will be collected at baseline, four weeks, and eight weeks to determine the efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* English speaking
* Literacy 6th grade and above
* Willingness to share contact information (home address, phone number)
* No current mindfulness practice
* Greenville residents or persons who are patients of the partnering organizations in the investigator's study.
* Self-reported physical activity level below the CDC recommended guidelines (150 minutes (2 hours and 30 minutes) a week of moderate-intensity, or 75 minutes (1 hour and 15 minutes ) a week of vigorous-intensity aerobic activity, or an equivalence combination of moderate- and vigorous intensity aerobic activity

Exclusion Criteria:

* <18 years old
* Non-English-speaking
* Literacy lower than 6th grade
* Inability to attend intervention sessions
* Already completed or attending a mindfulness-based intervention
* Current pregnancy
* Current/past psychosis
* Acute episode of a substance use disorder (past two weeks)
* Acute episode of depression in the past two weeks
* Moderate to severe traumatic brain injury or brain damage
* Persistent antisocial behavior
* Persistent self-injury requiring clinical management
* Unable to engage for physical or practical reasons (e.g., disabling physical problems, unable to comprehend material)
* Dementia
* Suicidality
* Inability to do light walking for 10 mins at a stretch
* Severely obese BMI (>50 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | Scale administered at pre-intervention (baseline), 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  Rapid Assessment of Physical Activity Scale: self-report scale of physical activity, with total score ranging from 1-10; higher scores indicate increased activity
Change in muscle strength | Assessment administered at pre-intervention (baseline), 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  Upper and lower muscle strength will be measured with the 30-second arm curl test (number of biceps curls completed while holding a hand weight of 2.27 kg for women and 3.63 kg for men) and the 30-second chair-stand test (Prakhinkit et al. 2014).
Change in sleep quality | Assessment administered at pre-intervention/baseline, 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  Pittsburgh Sleep Quality Index: 19 item self-report measure assessing sleep quality over the past month, total score ranging from 0 to 21, with higher scores indicating worse sleep quality
Change in flexibility | Assessment administered at pre-intervention (baseline), 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  The back scratch flexibility test (how close the hands can be brought together behind the back) and the chair sit-and-reach test will be used to measure upper and lower limb flexibility, respectively (Prakhinkit et al. 2014).
Change in agility | Assessment administered at pre-intervention (baseline), 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  The timed up-and-go test will be used as a measure of agility (Prakhinkit et al. 2014)
Change in dynamic balance | Assessment administered at pre-intervention (baseline), 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  The Star Excursion Balance Test will measure dynamic balance (Gribble, Hertel, and Plisky 2012)
Change in cardiorespiratory endurance | Assessment administered at pre-intervention (baseline), 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  6 minute walk test, measure includes how many meters the individual walks in 6 minutes around a 50-yard course (Prakhinkit et al. 2014)

SECONDARY OUTCOMES:
Change in perceived stress | Assessment administered at pre-intervention/baseline, 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  Perceived Stress Scale: 4 item self-report measure assessing perceived stress over the past month, total score ranges from 4 to 20, higher levels indicating higher levels of stress
Change in adherence to medications | Assessment administered at pre-intervention (baseline), 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  Adherence to Refills and Medications Scale: 12 item self-report scale assesses adherence to other medication treatments; scores range from 12-34, where lower scores indicate better adherence (adherence to medications not given as part of this study) (Kripalani et al. 2009)
Change in mindfulness skills | Assessment administered at pre-intervention (baseline), 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  The Five Facet Mindfulness Questionnaire: 39 self-report items assessing five dimensions of mindfulness. Items are rated on a 5 point scale ranging from 1 to 5, with total score ranging from 39 to 195. Higher scores indicate greater dispositional tendency to be mindful in daily life (e.g., observing, describing, acting with awareness, nonjudging of inner experience, nonreactivity to inner experiences).
Change in executive functioning | Assessment administered at pre-intervention (baseline), 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  Executive Function Index: A 27-item self-report inventory assessing five facets of executive functioning (Spinella, 2005); Items rated "how well the following statement describes me" 1 (not at all) to 5 (very much), range 27-135 with higher scores indicating higher levels of executive functioning.
Mindfulness practice behavior | Assessment administered at 4 weeks (post-intervention for experimental group), 8 weeks (post-intervention for control group and follow-up for experimental group)
  Additional mindfulness practices engaged in outside of the study sessions over the past month, assessed with four self-report items: 'Did you engage in mindfulness meditation in the past month?', 'How many days per week did you engage in mindfulness meditation?', 'How long in minutes did you meditate per session of mindfulness meditation?', 'Describe your practice of mindfulness meditation (what exercises/activities/techniques did you practice?)

OTHER OUTCOMES:
Demographic Information | Assessed at pre-intervention/baseline
  Age, race, ethnicity, marital status, language spoken, highest level of education, employment status, annual household income, health insurance, current smoking
Satisfaction with treatment | Administered at 4 weeks for experimental group and 8 weeks for control group.
  Treatment Satisfaction Survey (Zgierska et al. 2008), 5 item self-report measure, qualitative and quantitative items with quantitative scale ranging from 0 to 16, with higher scores indicating greater satisfaction with mindfulness intervention
Adverse childhood experiences | First 18 years of life
  Adverse Childhood Experiences Questionnaire: 10 item self-report scale assesses adverse events in the first 18 years of life (Felitti, 1998). Scores range from 0 to 10, with higher scores indicating greater number or adverse events.
Traumatic event history | Assessed at pre-intervention/baseline
  Life Events Checklist for DSM-5: 17 self-report items that assess a number of different types of traumatic events across the lifespan and personal occurrence versus learning about a traumatic event (Weathers et al., 2013). There is no formal scoring protocol, although endorsing 1 or more items indicates lifetime exposure to a traumatic event.
Use of psychological services | Assessed at pre-intervention/baseline
  The Adult Service Use Schedule: Fifteen open-ended, self-report items assessing use of psychological services, accessibility, and length of service use (Bower et al., 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Lu Shi, PhD, Principal Investigator — Clemson University
Locations (3):
- United States (3):
  - Clemson University, Clemson, South Carolina
  - Caine Halter Family YMCA, Greenville, South Carolina
  - Prisma Health-Upstate Internal Medicine Clinic, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside the research team